CLINICAL TRIAL: NCT01987284
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over, Multi-center Study Assessing the Safety, Tolerability and Efficacy of SER100 10 mg s.c. Twice Daily for 2 Days in Patients With Isolated Systolic Hypertension Insufficiently Treated With One or More Anti-hypertensives.
Brief Title: SER100 in Isolated Systolic Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Serodus AS (Industry)
Collaborators: Smerud Medical Research International AS (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-2271; 2013-001227-40 (EudraCT Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Isolated Systolic Hypertension
MeSH Terms: conditions — Isolated Systolic Hypertension | interventions — ZP120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SER100 (Experimental): SER100 10 mg s.c. twice daily
  Interventions: Drug: SER100; Drug: Placebo
- Placebo (Placebo Comparator): Placebo administered s.c. twice daily
  Interventions: Drug: SER100; Drug: Placebo

INTERVENTIONS:
Drug: SER100
Drug: Placebo

SUMMARY:
Isolated Systolic Hypertension (ISH)is the dominating hypertensive disease in elderly people. Much attention has recently been drawn to the strong relationship between the systolic blood pressure and cardiovascular morbidity.

In previous clinical studies carried out in individuals with normal blood pressure at baseline SER100 decreased primarily the systolic blood pressure. It is hypothesized that the effect on systolic blood pressure in hypertensive patients will be larger or equal to the fall seen in normotensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Mean systolic blood pressure ≥ 150 mmHg and mean diastolic blood pressure < 90 mmHg - as determined by daytime continuous ambulatory blood pressure measurement (ABPM)
* Male or female
* Age 50-80 years (both inclusive) at screening
* Patients must be on stable doses with one or more antihypertensives
* BMI <32 kg/m2
* Written informed consent

Exclusion Criteria:

* Acute myocardial infarction in the last 6 months before screening
* Stroke in the last 6 months before screening
* Uncompensated heart failure (NYHA Class IV)
* Angina pectoris with an anticipated need for administration of short-acting nitrates
* Known, severe sleep apnoea
* Abnormal laboratory values (i.e. > 2 x upper normal limit) at screening
* Subjects working night shifts (11 PM to 7 AM)
* Participation in any other clinical trial with an investigational medicinal product or device within 1 month prior to randomisation.
* Subjects with upper arm circumference ≤24 cm or ≥ 42 cm.
* Any general condition, serious disease or current evidence of any mental or physical disorder or collaboration attitude (e.g. dementia, substance abuse) which, in the judgment of the investigator makes the subject unsuitable for enrollment, and/or may interfere with the study evaluations or affect subject's safety and/or may cause risk for poor protocol compliance
* Pregnant or lactating women.
* Female subjects of childbearing potential, or male subjects whose female partner (unless post-menopausal for 1 year or surgically sterile) is unwilling to use adequate contraceptive measures throughout the duration of the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 4 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helga Gudmundsdottir, MD, Principal Investigator — Oslo University Hospital
Locations (7):
- Finland (2):
  - FinnMedi Oy/Valkeakoski District Hospital, Tampere
  - CRST/Turku University Hospital, Turku
- Semmelweiss University Hospital, Budapest, Hungary
- Norway (2):
  - Medi3 Innlandet, Hamar
  - Ulleval University Hospital, Oslo
- United Kingdom (2):
  - Northwick Park Hospital, Harrow, Middlesex
  - Brighton and Sussex University Hospital, Brighton